CLINICAL TRIAL: NCT06822673
Title: Impact of Mindfulness-Based Intervention on Biopsychosocial Factors Associated With Quality of Life in Children With Primary Headaches: A Randomized Controlled Trial
Brief Title: Impact of MBI on Biopsychosocial Factors and QOL in Children With Primary Headaches
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fatima Jinnah Women University (Other)
Responsible Party: Principal Investigator, Sadia Sohail, Researcher/Student, Fatima Jinnah Women University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FJWU/EC/2024/95; FJWU/EC/2024/95 (Other: Fatima Jinnah Women University)
Record Dates: First submitted 2025-01-23; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Primary Headache; Psychological Distress; Emotion Regulation; Childhood Trauma; Sedentary Behaviors; Mindfulness; Health-Related Quality-of-Life
Keywords: Pediatric Primary Headaches; Psychological Distress; Anxiety, Depression, Stress; Emotional Regulation; Childhood Trauma; Sedentary Behavior; Mindfulness-Based Intervention; Quality of Life; Randomized Controlled Trial; Headache Management; Non-Pharmacological Intervention
MeSH Terms: conditions — Emotional Regulation; Sedentary Behavior; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The interventional study model for this research follows a randomized controlled trial (RCT) design, which aims to evaluate the effectiveness of a Mindfulness-Based Intervention (MBI) in managing biopsychosocial factors associated with quality of life in children with primary headaches. Participants will be randomly assigned to either the intervention group, which will receive the MBI, or the control group, which will not receive any intervention. The study will adopt a pre-test, post-test, and follow-up assessment approach to measure changes in key variables, including psychological distress, emotion regulation, childhood traumatic experiences, sedentary behaviors, quality of life, mindfulness, and pediatric headache symptoms. The trial is currently in Phase 1, following the successful completion of pilot testing. At this stage, participants are being recruited for data collection.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Receiving Mindfulness Based Intervention) (Experimental): This arm includes children with primary headaches who will undergo the Mindfulness-Based Intervention (MBI). The intervention aims to improve biopsychosocial factors such as mindfulness, emotion regulation, psychological distress, and quality of life.
  Interventions: Behavioral: Mindfulness Based Intervention
- Control Group (No Intervention) (No Intervention): This arm consists of children with primary headaches who will not receive any intervention. This group will be used for comparison with Arm 1 to assess the effects of the MBI on biopsychosocial factors and quality of life. Participants in this arm will be assessed at the same time points.

INTERVENTIONS:
Behavioral: Mindfulness Based Intervention — The Mindfulness-Based Intervention will include techniques derived from the Mindfulness Matters Program protocol (for Children and Adolescents, 2019). It will consist of both formal and informal practices, which participants will engage in during sessions and at home. These practices will encompass body scan meditation, mindful eating, mindful sitting, walking exercises, attention-focusing activities, and more. The intervention will be delivered over eight weekly sessions, following a skill-building, educational approach.
  Arms: Interventional Group (Receiving Mindfulness Based Intervention)

SUMMARY:
* The Randomized Controlled Trial aims to evaluate the effectiveness of a Mindfulness-Based Intervention (MBI) in improving the quality of life and reducing psychological distress in children with primary headaches. This study focuses on children aged 8 to 12 years who experience primary headaches and aims to investigate the biopsychosocial factors influencing their well-being.
* The primary objectives of this study are:
* To assess the levels of mindfulness, emotional regulation, childhood traumatic experiences, psychological distress, and quality of life in children with and without primary headaches.
* To identify the key biopsychosocial factors that impact the quality of life in children experiencing primary headaches.
* To evaluate the effectiveness of mindfulness-based interventions in reducing psychological distress and enhancing the quality of life post-intervention.
* To compare the differences between the intervention and control groups regarding their biopsychosocial well-being before and after the intervention.
* To determine the long-term impact of the mindfulness-based intervention on psychological distress, quality of life, and headache frequency at a three-month follow-up.
* Participants in the study will be screened from an initial survey, based on those experiencing headaches and randomly assigned to intervention and control groups. The intervention group will undergo a structured mindfulness-based program, while the control group will receive standard care. Data will be collected at baseline, post-intervention, and during follow-up assessments to measure the intervention's impact.
* This study is significant as it aims to address the gaps in current research regarding pediatric primary headaches and their effect on psychological and social well-being. The findings may provide valuable insights for healthcare professionals to develop effective, non-pharmacological interventions to improve the quality of life of children suffering from primary headaches in Pakistan.

DETAILED DESCRIPTION:
Phases of the Study:

-Phase 1: Screening & Pre-Intervention Assessment Screening of children (ages 8-12) for primary headaches using standardized diagnostic criteria.

Assessment of biopsychosocial variables through validated psychological scales.

-Phase 2: Randomization & Intervention Random allocation of children into the intervention group, n=30 (receiving Mindfulness-Based Intervention) and control group, n=30 (receiving no intervention).

The intervention group would undergo an 8-week Mindfulness-Based Program, including techniques such as breathing exercises, guided imagery, body scanning, and mindful awareness practices.

-Phase 3: Post-Intervention Assessment Re-evaluation of all variables including psychological distress, mindfulness, and quality of life using the same assessment instruments.

Comparison of pre- and post-intervention outcomes.

-Phase 4: Follow-Up (3 Months Post-Intervention) Long-term impact assessment to determine sustained benefits of the intervention.

Ethical Considerations:

* Informed Consent: Parents/guardians will provide written consent before participation.
* Child Assent: Verbal and/or written assent will be obtained from children.
* Confidentiality: All data will be anonymized and securely stored.
* Right to Withdraw: Participants can leave the study at any point without any consequences.
* Free Psychological Support: Children in the intervention group will receive completely free mindfulness-based therapy sessions, and participation in these sessions is voluntary.
* After the study is completed, as an ethical and moral commitment, MBI therapy sessions would be offered to all those children also (who are willing) who were experiencing headaches but did not receive the intervention initially.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 to 12 years
* From an initial survey, those who experience headaches would be screened
* Children who are able to read and understand the English language, as the assessment instruments are in English, will be included.
* Both the children and their parents must consent to the child's participation in the study.

Exclusion Criteria:

* Children who are not students will be excluded from the study.
* Children with any diagnosed genetic disease or disorder, chronic disease, or disability will be excluded.
* Children with a current or past psychiatric disorder, especially those who have received treatment or medication for such conditions in the past year, will be excluded.
* Children who have been on any long-term medication for any disease or disorder will be excluded, as this may influence the results of the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality-of-Life | 10-12 weeks
  * Health-Related Quality of life refers to an individual's overall physical, social and emotional well-being related to health.
  * Measurement Tool: Pediatric Quality of Life Inventory (PedsQL)
  * Unit of Measure: Total score on PedsQL, with higher scores indicating better quality of life.
  * Detail: The PedsQL consists of multiple items assessing the impact of health conditions on a child's daily functioning. The scale evaluates the overall Health-Related Quality of life by aggregating responses across all items and domains. The total score is computed as the mean of all responded items.
Pediatric Headaches | 10-12 weeks
  * This outcome measure assesses the severity of headaches experienced by children.
  * Measurement Tool: Headache Screening Questionnaire (HSQ)
  * Unit of Measure: Total score, with higher values indicating greater headache severity.
  * Description: The HSQ consists of questions addressing headache related symptoms. This outcome would measure the changes in headache characteristics in response to MBI.
Mindfulness | 10-12 weeks
  * Mindfulness refers to the practice of present moment awareness.
  * Measurement Tool: Child and Adolescent Mindfulness Measure (CAMM)
  * Unit of Measure: Total CAMM score, with higher scores indicating greater mindfulness.
  * Detail: Mindfulness will be evaluated to determine whether MBI changes children's ability to focus on the present moment.

SECONDARY OUTCOMES:
Psychological Distress | 10-12 weeks
  * Psychological distress refers to the overall level of emotional discomfort or suffering experienced by an individual. It encompasses symptoms like anxiety, depression, and stress.
  * Measurement Tool: Depression Anxiety Stress Scales-Youth version (DASS-Y)
  * Unit of Measure: Total and subscale scores for depression, anxiety, and stress, with higher scores indicating greater distress.
  * Detail: The scale consists of 21 items, with seven items allocated to each of the three subscales: depression, anxiety, and stress. The overall aggregate score is then calculated to assess the individual's overall level of psychological distress.
  Psychological distress will be evaluated to determine the effectiveness of MBI related to emotional distress among children with primary headaches.
Emotion Regulation | 10-12 weeks
  * Emotion regulation refers to the ability to handle emotions effectively. This measure is crucial in assessing how children regulate emotions, particularly in relation to stressful or painful experiences like headaches.
  * Measurement Tool: Emotion Regulation Questionnaire for Children and Adolescents (ERQ-CA)
  * Unit of Measure: Total score, with higher scores indicating better emotion regulation abilities.
  * Detail: This measure assesses children's ability to manage emotions effectively.
Childhood Traumatic Experiences | 10-12 weeks
  * Childhood trauma includes adverse experiences such as abuse, neglect and other traumatic events.
  * Measurement Tool: Childhood Trauma Questionnaire-Short Form (CTQ-SF)
  * Unit of Measure: Total scores with higher scores indicating greater trauma exposure.
  * Detail: The scale assesses the cumulative impact of childhood traumatic experiences. The total score is used to evaluate the relationship between trauma exposure and primary headaches in children.
Sedentary Behaviors | 10-12 weeks
  * Sedentary behaviors involve prolonged inactivity with minimal physical movement.
  * Measurement Tool: International Physical Activity Questionnaire (IPAQ) Short Form
  * Unit of Measure: Average hours per day spent in sedentary activities.
  * Description: The study will assess the effect of MBI on sedentary behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Iram Gul, PhD, Study Chair — Fatima Jinnah Women University
Locations (1):
- Fatima Jinnah Women University, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data, including primary and secondary outcome measures, excluding personally identifiable information will be shared. IPD that underlie results in a publication will be shared in line with ethical considerations and confidentiality policies.
Supporting Information: SAP, CSR
Time Frame: The data will be available after study completion and publication of primary findings (tentatively from December, 2025) and will remain available for 1 year.
Access Criteria: * Qualified researchers affiliated with recognized academic institutions or research organizations with an approved data-sharing request will be able to access the IPD. Researchers may request access to summary findings and non-identifiable data under ethical and institutional guidelines.
  * They will be able to access de-identified IPD related to outcome measures.
  * Requests will be reviewed by the principal investigator and an ethics committee based on scientific merit and ethical considerations. Approved researchers must sign a data-sharing agreement outlining data use restrictions.
  * Data will be shared through a secure repository or institutional data-sharing platform, ensuring compliance with confidentiality and ethical standards.